CLINICAL TRIAL: NCT06212453
Title: Evaluation of the Functional Outcomes After Bilateral, 3D Ultrasound-guided Focal Thermal Ablation of the Prostate Transition Zone, in Patients with Benign Prostatic Hyperplasia-related Obstruction
Acronym: BETTANY
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP230759; 2023-A02267-38 (Other: ID-RCB)
Record Dates: First submitted 2023-11-24; First posted 2024-01-18 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Intervention Model Description: Targeted Microwave Ablation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- patients with BPH (Experimental): Targeted Microwave Ablation
  Interventions: Procedure: Targeted Microwave Ablation

INTERVENTIONS:
Procedure: Targeted Microwave Ablation — 3D ultrasound-guided focal thermal ablation of the prostate transition zone

SUMMARY:
The aim of the current study is to evaluate the efficacy of transperineal focal microwave ablation (TMA) of the prostate transition zone as a new treatment for lower urinary tract symptoms (LUTS) due to benign prostatic hyperplasia (BPH) within a prospective single-institutional pilot study.

DETAILED DESCRIPTION:
Transurethral resection of the prostate, laser vaporization or enucleation, and simple open prostatectomy represent the current gold standard surgical interventions for BPH-related obstruction. However, these treatments are burdened by their invasiveness, intra and post-operative morbidity, and long-term complications, including ejaculatory dysfunction (70%), urethral strictures (7%), urinary incontinence (2%), and bleeding. Laser-based surgical strategies have only partially overcome these drawbacks.

To provide a personalized therapy for the treatment of BPH related-symptoms, several minimally invasive surgical therapies (MISTs) were developed with the aim of achieving outcomes comparable to the gold standard invasive procedures while minimizing SD and other complications. Urolift implants and Rezum system have demonstrated less complication rate and hospitalization time than standard surgeries.

Recently, 3D ultrasound-guided transperineal focal microwave ablation (TMA) was developed as a focal treatment for localized prostate cancer. Ultrasound-MRI image fusion was performed with organ-based tracking-registration using KOELIS Trinity™ (Koelis, Meylan, France). Microwave thermal ablation was provided by the TATO generator (Biomedical Srl, Firenze, Italy) using a single 17G needle inserted transperineally. This treatment was reported to be safe, precise, and feasible in an outpatient setting.

ELIGIBILITY:
Inclusion Criteria:

* Man over 40 years old
* Indication of surgical management for BPH
* Prostate volume ≥30 cc and ≤100 cc as evaluated by ultrasonography
* IPSS score ≥15
* Qmax ≤12 ml/s
* Affiliated to the French national social security system
* Patient suitable for IV sedation or general anesthesia and focal microwave ablation
* Wish and able to comply with planned visits
* Able to express his consent
* Signed informed consent form

Exclusion Criteria:

* Unwillingness to accept the treatment
* Neurological pathology responsible for micturition disorders
* History of prostatic surgery
* History of prostatic arterial embolization
* Prostate protrusion Index of grade 2 (>5 mm) or more as evaluated by ultrasonography.
* Stenosis of the urethra
* History of prostate cancer
* History of radiotherapy or pelvic surgery
* Life expectancy <2 years
* Inability to understand the informed consent document, to give consent voluntarily or to complete the study tasks.
* Participation in another clinical study involving an investigational product within 1 month before study entry.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Difference between IPSS score at baseline and at 3 months | 3 months
  The International Prostate Symptom Score IPSS is a self-questionnaire - It contains seven questions about symptoms related to BPH and one question about the patient's perceived quality of life.
  The seven questions are scored from 0 to 5. The sum of the 7 items gives the International Prostate Symptom Score in terms of severity (out of 35):
  0-7 Mildly symptomatic - 8-19 Moderately symptomatic - 20-35 Severely symptomatic - Efficacy of the intervention with a decrease of at least 6 points on IPSS score between 3 months and baseline.

SECONDARY OUTCOMES:
Length of hospital stay | 1 month
Need for postoperative bladder catheterization | 1 month
Duration of postoperative bladder catheterization | 1 month
Postoperative pain | two hours after surgery
  Visual analogue scale (1 to 10)
Dimensions of transitional zone tissue ablation | 7 days
  Measurement on prostatic mpMRI performed at day 7
Male Sexual Health Questionnaire-ejaculatory dysfunction Short Form (MSHQ-EjD-SF) | 1, 3 and 12 months
  4 items to assess ejaculatory functions This score is based on 3 questions concerning symptoms (score from 1 to 15) and one question about discomfort (score from 0 to 5).
International Index of Erectile Function (IIEF-15) | 1, 3 and 12 months
  15 items to assess ejaculatory functions and global sexual life - This score is based on 3 questions concerning symptoms (score from 1 to 15) and one question about discomfort (score from 0 to 5).
IPSS score | 1, 3 and 12 months
  to assess urinary tract symptoms - 0-7 Mildly symptomatic 8-19 Moderately symptomatic 20-35 Severely symptomatic
Urinary Symptom Profile (USP) | 1, 3 and 12 months
  to assess urinary tract symptoms
Qmax | 1, 3 and 12 months
  to assess urinary tract symptoms
Patients perspectives and treatment preferences | Baseline
  Characterization of patient motivation to undergo TMA at baseline, as assessed by the patient perspective questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas BARRY DELONGCHAMPS, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Cochin, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yuan JQ, Mao C, Wong SY, Yang ZY, Fu XH, Dai XY, Tang JL. Comparative Effectiveness and Safety of Monodrug Therapies for Lower Urinary Tract Symptoms Associated With Benign Prostatic Hyperplasia: A Network Meta-analysis. Medicine (Baltimore). 2015 Jul;94(27):e974. doi: 10.1097/MD.0000000000000974. PMID 26166130
- [Background] Cornu JN, Ahyai S, Bachmann A, de la Rosette J, Gilling P, Gratzke C, McVary K, Novara G, Woo H, Madersbacher S. A Systematic Review and Meta-analysis of Functional Outcomes and Complications Following Transurethral Procedures for Lower Urinary Tract Symptoms Resulting from Benign Prostatic Obstruction: An Update. Eur Urol. 2015 Jun;67(6):1066-1096. doi: 10.1016/j.eururo.2014.06.017. Epub 2014 Jun 25. PMID 24972732
- [Background] McVary KT, Gange SN, Gittelman MC, Goldberg KA, Patel K, Shore ND, Levin RM, Rousseau M, Beahrs JR, Kaminetsky J, Cowan BE, Cantrill CH, Mynderse LA, Ulchaker JC, Larson TR, Dixon CM, Roehrborn CG. Minimally Invasive Prostate Convective Water Vapor Energy Ablation: A Multicenter, Randomized, Controlled Study for the Treatment of Lower Urinary Tract Symptoms Secondary to Benign Prostatic Hyperplasia. J Urol. 2016 May;195(5):1529-1538. doi: 10.1016/j.juro.2015.10.181. Epub 2015 Nov 22. PMID 26614889
- [Background] Oelke M, Bachmann A, Descazeaud A, Emberton M, Gravas S, Michel MC, N'dow J, Nordling J, de la Rosette JJ; European Association of Urology. EAU guidelines on the treatment and follow-up of non-neurogenic male lower urinary tract symptoms including benign prostatic obstruction. Eur Urol. 2013 Jul;64(1):118-40. doi: 10.1016/j.eururo.2013.03.004. Epub 2013 Mar 13. PMID 23541338
- [Background] Gratzke C, Bachmann A, Descazeaud A, Drake MJ, Madersbacher S, Mamoulakis C, Oelke M, Tikkinen KAO, Gravas S. EAU Guidelines on the Assessment of Non-neurogenic Male Lower Urinary Tract Symptoms including Benign Prostatic Obstruction. Eur Urol. 2015 Jun;67(6):1099-1109. doi: 10.1016/j.eururo.2014.12.038. Epub 2015 Jan 19. PMID 25613154
- [Background] Leonardo C, Lombardo R, Cindolo L, Antonelli A, Greco F, Porreca A, Veneziano D, Pastore A, Dalpiaz O, Ceruti C, Verze P, Borghesi M, Schiavina R, Falabella R, Minervini A; AGILE Group. What is the standard surgical approach to large volume BPE? Systematic review of existing randomized clinical trials. Minerva Urol Nefrol. 2020 Feb;72(1):22-29. doi: 10.23736/S0393-2249.19.03589-6. Epub 2019 Oct 10. PMID 31619035